CLINICAL TRIAL: NCT04857385
Title: Radial Artery Puncture Hemostasis: Physical, Biological and Chemical Methods
Brief Title: Radial Artery Puncture Hemostasis Study
Acronym: RAPHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Responsible Party: Principal Investigator, Istvan Edes, Associate Professor, Semmelweis University Heart and Vascular Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPHE-001
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Radial Artery Hemostasis
Keywords: Radial artery puncture; Radial artery occlusion; Radial artery bleeding
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Terumo TR Band (Active Comparator): Physical standard of care radial hemostasis device.
  Interventions: Device: Radial artery hemostasis
- StatSeal (Experimental): Potassium-ferrate based chemical hemostasis device.
  Interventions: Device: Radial artery hemostasis
- Axiostat (Experimental): Chitosan based biological hemostasis device.
  Interventions: Device: Radial artery hemostasis

INTERVENTIONS:
Device: Radial artery hemostasis — Each of the devices will be assessed for radial artery hemostasis.

SUMMARY:
RAPHE is an open label randomized clinical trial to assess physical, biological and chemical methods of radial artery puncture hemostasis following coronary catheterization.

A total of 600 subjects will be randomized in a 1:1:1 fashion to either the StatSeal, Axiostat or TR Band hemostasis devices.

Follow-up of the subject will take place 60 days after the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiogram planned from a radial artery approach
* Use of 5, 6 or 7 French sheaths

Exclusion Criteria:

* Radial artery diameter <1.8 mm as measured via ultrasound
* Established peripheral arterial disease
* Known autoimmune illness
* Hemodynamic instability
* Pregnant or nursing
* Condition following resuscitation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion | 24 hours post-procedure or at hospital discharge (whichever comes first)
  Frequency of radial artery occlusion after hemostasis
Radial artery occlusion | 60 days (+/-10 days) post-procedure
  Frequency of radial artery occlusion after hemostasis
Radial artery (pseudo)aneurysm formation | 24 hours post-procedure or at hospital discharge (whichever comes first)
  Frequency of radial artery (pseudo)aneurysm formation after hemostasis
Radial artery (pseudo)aneurysm formation | 60 days (+/-10 days) post-procedure
  Frequency of radial artery (pseudo)aneurysm formation after hemostasis
Radial artery fistula formation | 24 hours post-procedure or at hospital discharge (whichever comes first)
  Frequency of radial artery arteriovenous fistula formation after hemostasis
Radial artery fistula formation | 60 days (+/-10 days) post-procedure
  Frequency of radial artery arteriovenous fistula formation after hemostasis
Radial artery bleeding | 24 hours post-procedure or at hospital discharge (whichever comes first)
  Bleeding from the radial artery puncture, classified via the EASY method
Radial artery bleeding | 60 days (+/-10 days) post-procedure
  Bleeding from the radial artery puncture, classified via the EASY method

SECONDARY OUTCOMES:
Initial compression time of hemostatsis device | Up to 30 minutes post-procedure
  Initial time (in minutes) of the hemostasis device, needed to achieve primary patent hemostasis
Overall compression time | Up to 24 hours post-procedure
  Overall time (in minutes) of device use as a hemostatis tool
Number of compression devices needed | Up to 24 hours post-procedure
  Overall number of compression devices needed for hemostatis

OTHER OUTCOMES:
Need for bail-out device | Up to 24 hours post-procedure
  Percentage of patients requiring bail-out hemostasis devices

CONTACTS AND LOCATIONS:
Overall Officials: István F Édes, MD PhD, Principal Investigator — Semmelweis Univeristy Heart and Vascular Center
Locations (3):
- Hungary (3):
  - University of Szeged, Department of Invasive Cardiology, Szeged, Csongád-Csanád
  - Department of Cardiology and Cardiac Surgery, Debrecen, Hajdú-Bihar
  - Semmelweis University Heart and Vascular Center, Budapest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kulyassa P, Nemeth BT, Ehrenberger R, Ruzsa Z, Szuk T, Fehervari P, Engh MA, Becker D, Merkely B, Edes IF. The Design and Feasibility of the: Radial Artery Puncture Hemostasis Evaluation - RAPHE Study, a Prospective, Randomized, Multicenter Clinical Trial. Front Cardiovasc Med. 2022 May 27;9:881266. doi: 10.3389/fcvm.2022.881266. eCollection 2022. PMID 35694680